CLINICAL TRIAL: NCT07068971
Title: Assessing the Feasibility of a Multi-modal Intervention for Sleep Disturbances in Patients With Advanced Cancer
Brief Title: Sleep Well At Night
Acronym: SWAN
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Our Lady's Hospice and Care Services (Other)
Collaborators: St Vincent's University Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Prof Andrew Davies, Professor of Palliative Medicine, Our Lady's Hospice and Care Services
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RS23-076; RS23-076 (Other: St Vincent's University Hospital)
Record Dates: First submitted 2025-06-26; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Sleep Disturbance in Advanced Cancer
Keywords: Non-pharmacological; Multimodal; Interventional; Feasibility study; Advanced cancer
MeSH Terms: interventions — Ultraviolet Therapy; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Receiving intervention (Experimental): Participants recruited to the study will receive the multimodal intervention as described.
  Interventions: Behavioral: Online cognitive behavioural therapy for insomnia, bright light therapy, activity

INTERVENTIONS:
Behavioral: Online cognitive behavioural therapy for insomnia, bright light therapy, activity — Multimodal intervention

SUMMARY:
Research has shown that the incidence of sleep disturbances in people with cancer is much higher than in the general population. Sleep problems can lead to worse symptoms, quality of life, and potentially impact outcomes. The most common treatment of sleep disturbances is medication which often comes with unwanted side-effects and risk. This study aims to test whether a non-drug intervention can be given to people with cancer to help with sleep disturbances.

The study will take place over 8-weeks. The first and final week of the study involves assessments (further described below) while the intervention will take place over weeks 2-7. The intervention involves an online cognitive behavioural therapy course, daily bright light therapy and engaging with an activity plan.

The initial review aims to identify any reversible causes of the sleep disturbance, including reviewing uncontrolled symptoms and medications.

Cognitive behavioural therapy for insomnia (CBT-I) has been shown to be effective at improving the time it takes for people to fall asleep and reducing the amount of time you wake up in the night.

Light therapy mimics our natural exposure to sunlight. Light exposure may help to improve sleep during the night, mood, and activity or attention levels during the day.

Physical activity levels will also be reviewed. Interests and barriers to activity will be discussed and goals will be set for activity. This will be reviewed weekly.

Questionnaires will be completed in the first and final week of the study to assess sleep, symptoms and quality of life. Wrist actigraphy, thigh accelerometry and a sleep diary will also be used on the first and final week of the study to assess sleep, activity and subjective sleep patterns.

DETAILED DESCRIPTION:
Advances in cancer treatments have improved prognosis for many patients, placing a heightened demand on clinical care to provide quality of life as well as quantity of life. Individuals with advanced cancer face progressive symptoms that are a major source of suffering and impairment. Sleep disturbance is a prevalent, but often overlooked symptom, affecting up to 96% of patients with advanced cancer. While there are multiple types of sleep disorders affecting patients with advanced cancer, insomnia seems to be the most prevalent sleep disorder in this patient cohort, occurring at various points in the patient's disease and treatment trajectory. Adequate sleep is essential for maintaining normal function and overall existence. Inadequate sleep may further compound illness and impair recovery. Sleep disturbances are associated with fatigue, accidents/injuries, anxiety and depression, cognitive impairment and delirium and immunosuppression. In addition, sleep disturbance is associated with aberrant patterns of cortisol secretion, which can impair the cellular immunity responsible for mounting a defence against tumours. Pharmacotherapy is the most common treatment for sleep disturbances, despite the numerous associated adverse effects and absence of empirical evidence of their efficacy and innocuity in this patient population. Multiple studies have recognised that patients with advanced cancer are at an increased risk of harm induced by medications due to age, polypharmacy and co-morbidities that can alter pharmacodynamics. Yet, despite the evidence of harmful effects of hypnotics and the lack of evidence to support their use, they are routinely prescribed as first-line treatment for the management of sleep disturbances in patients with advanced cancer.

Cognitive behavioural therapy for insomnia (CBT-I) is considered the non-pharmacological first-line treatment to manage insomnia in adults. CBT for insomnia includes various components that helps the patient to learn coping skills and ways to prevent or mitigate the severity of future episodes.

Both bright white light therapy and exercise have proven to be successful non-pharmacological methods of optimising daytime activity, improving sleep duration and enhancing symptoms and quality of life in patients with cancer.

Study interventions

1. CBT-I is a first-line treatment for insomnia. The online course consists of four CBT-I sessions and allows the individual to complete one module per week in the comfort of their own home. Online CBT-I has been shown to be as effective as face-to-face CBTI. CBT-I covers cognitive and behavioural aspects to understand sleep processes and improve sleep duration and quality.
2. Bright light therapy has been shown to be effective at improving night-time sleep and daytime physical activity. It is delivered from a light box. The participants will be advised to sit near the light box for 30 minutes each morning. Participants can continue with other activities, such as eating breakfast, whilst sitting with the light box.
3. An individualised physical activity plan will be created to encourage increased daytime physical activity and reduced daytime sedentary behaviour. Existing physical activity levels will be considered, any barriers to physical activity addressed, and goals for physical activity set. These will be reviewed on a weekly basis and adjusted as appropriate. For example, if goals are easily being achieved, further activity increases will be advised. If the patient struggles to meet goals, their goal will be lowered. Patients will be provided with a generic watch activity tracker to help them to monitor their progress.

Study Duration/ Study Timeline:

All participants will receive the intervention over an 8-week period. Where possible, participants baseline and repeat assessments will be arranged to avoid assessments taking place during a week of intravenous systemic anticancer therapy as this may impact symptoms and results.

At baseline, participants will complete three questionnaires related to symptoms, sleep disturbance and quality of life. Participants will be given a Polar Unite watch to wear for the duration of the study (8 weeks) as a primary objective measure for the purpose of measuring sleep and activity. Participants will also complete a sleep diary during the first week and wear a thigh accelerometer as a secondary objective outcome to measure activity including time spent lying, sitting, standing and stepping.

At the end of week one, participants will return the sleep diary and thigh accelerometer and they will be provided with and educated on the use of the bright white light box and the CBT-I platform. An individualised activity plan will be created between the research team and the participant. Participants will receive 6 weeks of the intervention prior to a final week where they repeat the questionnaires, thigh accelerometer and diary completion. Weekly virtual contacts will take place throughout the intervention. These will consider adverse events, technical complications, to advise on adjustments to the activity plan and to encourage engagement with the intervention.

Baseline - beginning of week one Participants will attend to meet the researcher at a convenient location. The initial clinical review is expected to take approximately 60 minutes. A checklist will be used throughout to ensure all steps are completed. The participant will be provided with a Polar Unite watch, a thigh accelerometery device and a sleep diary. The participant will wear the Polar Unite watch for the duration of the study (8 weeks). They will wear the thigh accelerometer device for 3 days and 3 nights (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays) of the first week to capture their baseline activity and for 3 days and 3 nights (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays) of the final week (post-intervention). The thigh accelerometer and sleep diary will be returned/collected on Friday (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays) of the same week and at this point the patient will begin to receive the intervention (CBT-I, bright white light therapy and their activity plan).

The baseline assessment may highlight physical/psychological symptoms abnormalities. In this event, and with the patient's verbal consent, the clinical team (GP, oncologist, palliative physician) will be made aware of the findings to review further.

The consent form and baseline assessments will be completed to include:

1. Demographics: Age, sex, race, living situation, bedroom situation, sleep posture.
2. Clinical history: cancer history (date of diagnosis, type of cancer, stage of cancer and current oncology treatment, past medical history, medication).
3. Lifestyle: smoking history, caffeinated drink use, alcohol use, daily activity.
4. The following assessment tools; PSQI MSAS-SF EORTC QLQ-C15-PAL Dreams & Nightmares Questionnaire

End of week one The researcher will meet with the participant again on Friday of week one (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays). This meeting will focus on an introduction to the interventions and the rationale behind them, including CBT-I and bright white light therapy. It will also involve a discussion around personal interests, barriers to activity, and goals to improve activity levels throughout the day.

Weeks 2-7 - Ongoing intervention Virtual contacts will occur over the phone. The research team will assess for any technical challenges. Goals will be recalled and engagement in the intervention encouraged and any barriers will be addressed.

Week 8 - Completion of intervention and repeat monitoring The researcher will meet with the participant on Monday (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays) and repeat the assessment tools (PSQI, MSAS-SF, EORTC QLQ-C15-PAL). The thigh accelerometer and sleep diary will be repeated again for 3 days and 3 nights and returned/collected on the Friday (+/- 3 days and 3 nights to allow for flexibility in the case of clashing appointments/bank holidays).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years old and over
2. Diagnosis of advanced cancer (locally advanced, metastatic)
3. Subjective sleep disturbance
4. Total score of 5 or more on PSQI
5. Eastern Cooperative Oncology Group (ECOG) performance status 1-3
6. Attending outpatients (oncology and/or palliative care)
7. Estimated prognosis of > 3 months

Exclusion Criteria:

1. Inpatient
2. ECOG performance status 4
3. Cognitive impairment limiting the ability to complete assessment tools and sleep diary
4. Engaged in shift work
5. A recent exacerbation of symptoms (e.g. pain/nausea/dyspnoea) which may impact sleep
6. History of uncontrolled mania or bipolar disorder
7. Recent history or current thoughts of self-harm or suicide
8. Recent change in antidepressant medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-08-24 (Estimated); Study Completion 2025-08-24 (Estimated)

PRIMARY OUTCOMES:
Retention rate | through study completion - 8 weeks
  considering the number of patients who entered the study and completed the study.
Recruitment | one year
  considering the number of patients approached to take part in the study who then entered the study
Completion of the intervention | 8 weeks
  Considering engagement with various interventions. The case report form will capture engagement with online cognitive behavioural therapy for insomnia where progress can be viewed online and the sleep diary will be reviewed. The participant will report on use of the bright light therapy box and activity levels throughout the study.
Acceptability | 8 weeks
  A patient acceptability questionnaire of various aspects of the study, including interventions and study protocol, will be completed at the end of the study.

SECONDARY OUTCOMES:
Sleep quality | Week 8
  Using brief Pittsburgh Sleep Quality Index. A score of 5 or more indicates poor sleep question. Maximum score of 21. The higher the score, the poorer the sleep quality.
Physical symptoms | Week 8
  Assessed using the Memorial Symptom Assessment Scale-Short Form. This is a 32-item tool, is a valid and reliable tool within the cancer population for assessing physical and psychological symptoms over the preceding week. Each symptom is only rated if present. This tool provides sub-scale scores rather than a total score. No "maximum score" is reported - rather average subscale scores. The higher the mean, the greater the symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Professor Andrew Davies, Principal Investigator — Our Lady's Hospice & Care Services
Locations (1):
- Our Lady's Hospice & Care Services, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study, and thus is not sufficiently powered to provide robust evidence of the efficacy of the intervention.
  Data from a future definitive study will be shared with bona fide researchers subject to them signing a data sharing agreement.